CLINICAL TRIAL: NCT01127620
Title: A Phase III, Comparative Study for the Efficacy and Safety of Bilastine 20 mg Versus Cetirizine 10 mg and Placebo in the Treatment of Perennial Allergic Rhinitis During 4 Weeks, Followed by a Long-term Safety Extension With Bilastine 20 mg
Brief Title: Efficacy Study for the Symptomatic Treatment of Perennial Allergic Rhinitis With a 1 Year Safety Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BILA 1503/RAP
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Allergic Rhinoconjunctivitis; Persistent allergic rhinitis; Hay fever; Allergic Rhinitis; Sneezing; Nasal congestion; Rhinorrhea; Nasal itching; Ocular itching; Ocular tearing; Antihistamine
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic; Sneezing; Nasal Obstruction; Rhinorrhea | interventions — bilastine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bilastine (Experimental): 20 mg encapsulated tablets
  Interventions: Drug: Bilastine
- Cetirizine (Active Comparator): 10 mg encapsulated tablets
  Interventions: Drug: Cetirizine
- Placebo (Placebo Comparator): Encapsulated tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bilastine — 20 mg encapsulated tablets
  Arms: Bilastine
Drug: Cetirizine — 10 mg encapsulated tablets
  Other Names: Zyrtec
  Arms: Cetirizine
Drug: Placebo — encapsulated tablets
  Arms: Placebo

SUMMARY:
Double-blind phase: The objective of the study was to evaluate the efficacy and safety of Bilastine 20 mg, compared to Cetirizine and placebo for the treatment of perennial allergic rhinitis.

Open-label Phase: The objective of this extension was to evaluate the long-term safety of Bilastine 20 mg during one year in the symptomatic treatment of perennial allergic rhinitis

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled, parallel-group, international, multicenter study followed by an open label extension. Duration of the double-blind period was 28 days and the duration of the open label period was 12 additional months.

The primary efficacy variable of the double-blind period was the area under curve (AUC) of total symptoms scale (TSS) from baseline (defined as the mean of 6 last points of the patients' diary before randomization) to D28 visit according to the patient's assessment on reflective symptoms. 650 patients were included in the study and 614 completed the double-blind phase. Out of the 614 patients who completed the double blind period, a total of 513 patients started the open label period with Bilastine 20 mg (83.6%)

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged from 12 to 70 years of age
* Patients with a documented clinical history of PAR for at least 2 years prior to the study inclusion
* Positive skin prick test for at least one of the following perennial allergens (house-dust mites, Dermatophagoides pteronyssinus or D. farinae, animal danders, dogs or cats, molds, etc.)
* Patients had to have a sum in the previous 6 assessments of the reflective nasal symptoms score equal to or greater than 30 (≥30 over 72). Additionally, at the time of randomization patients had to have positive symptomatology in instantaneous nasal symptoms equal or greater than 5 (≥5 over 12).
* Women of childbearing potential had to have a negative pregnancy test and had to use an effective contraceptive method.
* Provision of written informed consent to participate and willing to attend the required visits scheduled in the protocol
* The criteria to continue with the open label period included previous participation in the double blind period, eligibility for a long-term symptomatic treatment according to the investigator assessment and patient willingness to follow the treatment for one year.

Exclusion Criteria:

* Patients who have non-allergic rhinitis (vasomotor, infectious, drug-induced, etc.).
* Negative skin prick test (as defined in point 6.1.1.).
* Patients with nasal polyps or a significant deviation of the nasal septum as judged by the investigator as well as nasal intervention in the previous 6 months.
* Any other nasal illness that can interfere with the aim of the study.
* Patients who have acute or chronic sinusitis as judged by the investigator.
* Patients who are also diagnosed with SAR (seasonal allergic rhinitis), and the inclusion and follow-up during the double-blind phase in this study is concurrent with the pollen season.
* Immunotherapy (6 months): In case of patients under immunotherapy the treatment had to have started more than 6 months prior to the start of the study, the doses could not be modified during the study, and any doses could not be administered 24 hours before any study visit..
* Patients who are taking or have taken specified medications prior to randomisation in the study and have not complied with the specified washout period
* Severe concomitant disease that could interfere with treatment response (hepatic, renal, cardiovascular), electrocardiographic abnormalities, arrhythmia, recent acute myocardial infarction or neoplastic diseases

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Double-blind phase: AUC of TSS throughout the study | 28 days
  Area under curve (AUC) of total symptoms scale (TSS) from baseline (defined as the mean of 6 last points of the patients' diary before randomization) to D28 visit according to the patient's assessment on reflective symptoms.
Open-label phase: Long-term safety | 12 months
  Evaluation of the long-term safety of Bilastine 20 mg during one year in the symptomatic treatment of perennial allergic rhinitis. The tolerability of the study drug was assessed by means of: Adverse events (comparing the profiles throughout the course of the study), ECGs on M3, M6, M9 and M12 visits and routine laboratory analyses (haematology and biochemistry) performed at M3, M6, M9 and M12 visits.

SECONDARY OUTCOMES:
AUC of TSS since baseline to D28 according to the patient's assessment on instantaneous symptoms. | 28 days
Change in the TSS on D14 and D28 visits versus D0 visit according to the patient and investigator's assessments (at the moment of the visits) | Day 14 and day 28
Change in Nasal Symptoms Score (NSS) | Day 14 and day 28
  Change in Nasal Symptoms Score (NSS) on symptoms scale on D14 and D28 visits versus D0 visit according to the patient and investigator's assessment (at the moment of the visits)
Change in Non Nasal Symptoms Score (NNSS) | Day 14 and day 28
  Change in Non Nasal Symptoms Score (NNSS) on symptom scale on D14 and D28 visits versus D0 visit according to the patient and investigator's assessment (at the moment of the visits)
Change in individual nasal and non nasal symptoms | Day 14 and day 28
  Change in each of the NSS or NNSS on symptoms scale on D14 and D28 visits versus D0 visit according to the patient and investigator's assessments (at the moment of the visits)
AUC of NSS, NNSS and each individual nasal andn non nasal symptom | 28 days
  AUC of NSS, NNSS and each of the nasal and non nasal symptoms scores on symptoms scale from baseline to D28, according to the patient's assessment on reflective symptoms
AUC of NSS, NNSS and each individual symptom according to patient's instantaneous assessment | 28 days
  AUC of NSS, NNSS and each of the nasal and non nasal symptoms scores on symptoms scale from baseline to D28, according to the patient's assessment on instantaneous symptoms. Time to maximum relief of symptoms
Overall assessment of discomfort | Day 14 and day 28
  Overall assessment of discomfort caused by allergic rhinitis using a visual analog scale (VAS) on D14 and D28 visits
Investigator's clinical global impression | 28 days
Quality of Life change from baseline | 28 days
Responders rate | 28 days
  Responders were classified based on their total symptom score decrease to baseline: <25%, 25%-50%, 50%-75%, >75% and were described by treatment group with their percentage and 95% confidence interval.
Time to maximum response | 48 hours
  Time to maximum response was described using Kaplan-Meier estimates and was compared (Log-rank test) between treatment groups.
Safety and tolerability | 28 days
  The tolerability of the study drug was assessed by means of: Adverse events (comparing the profiles throughout the course of the study, ECGs on D0 and D28 visits and routine laboratory analyses (haematology and biochemistry) performed at D0 and D28 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Prof. MD., Principal Investigator — Barlicki University Hospital, Medical University of Lodz (Poland)

REFERENCES:
- [Background] Bousquet J, Ansotegui I, Canonica GW, Zuberbier T, Baena-Cagnani CE, Bachert C, Cruz AA, Gonzalez SN, Kuna P, Morais-Almeida M, Mullol J, Ryan DP, Sanchez-Borges M, Valiente R, Church MK. Establishing the place in therapy of bilastine in the treatment of allergic rhinitis according to ARIA: evidence review. Curr Med Res Opin. 2012 Jan;28(1):131-9. doi: 10.1185/03007995.2011.648263. Epub 2011 Dec 22. PMID 22149770
- [Result] Sastre J, Mullol J, Valero A, Valiente R; Bilastine Study Group. Efficacy and safety of bilastine 20 mg compared with cetirizine 10 mg and placebo in the treatment of perennial allergic rhinitis. Curr Med Res Opin. 2012 Jan;28(1):121-30. doi: 10.1185/03007995.2011.640667. Epub 2011 Nov 30. PMID 22077106